CLINICAL TRIAL: NCT01603173
Title: A Randomized, Open Label, Two-Treatment, Two-Period, Two-Sequence, Crossover, Single Dose, Bioequivalence Study of Quetiapine Fumarate Tablets 25 mg With Seroquel® 25 mg in Normal, Healthy, Adult, Human Subjects, Under Fasting Condition
Brief Title: Bioequivalence Study of Quetiapine Fumarate Tablets 25 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/ARL/233
Record Dates: First submitted 2012-04-19; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Fasting State
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine Fumarate Tablets 25 mg (Experimental): Quetiapine Fumarate Tablets 25 mg of M/s Ipca Laboratories Limited, India
  Interventions: Drug: Quetiapine Fumarate Tablets 25 mg
- Seroquel® (Active Comparator): Seroquel® (Quetiapine Fumarate) Tablets 25 mg of M/s AstraZeneca Pharmaceuticals LP, USA
  Interventions: Drug: Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate Tablets 25 mg — 25 mg tablet once a day
  Other Names: Test Product
  Arms: Quetiapine Fumarate Tablets 25 mg
Drug: Quetiapine Fumarate — 25 mg tablet once a day
  Other Names: Seroquel®
  Arms: Seroquel®

SUMMARY:
This is a randomized, open Label, two-treatment, two-period, two-sequence, crossover, single dose pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fasting condition in normal, healthy, adult, human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Quetiapine Fumarate Tablets 25 mg of M/s Ipca Laboratories Limited, India and the corresponding Reference Product: Seroquel® (Quetiapine fumarate) Tablets 25 mg of M/s AstraZeneca Pharmaceuticals LP, USA, under fasting condition in normal, healthy, adult, human subjects in a randomized crossover study.

The study was conducted with 54 healthy adult subjects. In each study period, a single 25 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 11 days including washout period of at least 7 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female human subjects, age in the range of 25 - 45 years and weight ≥60 kg.
2. BMI within range of 18.5kg/m2 - 30 kg/m2.
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and oral temperature).
4. Subjects with blood pressure more than or equal to 110/70mmHg at the time of screening and at the time of check in for each study period.
5. Subjects with clinically acceptable findings as determined by haemogram, biochemistry, serology (HIV, Hepatitis B and Hepatitis C), urinalysis, 12 lead ECG and chest X-ray (chest X-ray if required).
6. Willingness to follow the protocol requirements as evidenced by written informed consent.
7. Confirming and agreeing to, not using any prescription and over the counter medications including vitamins and minerals for 14 days prior to study and during the course of the study.
8. No history of drug abuse in the past one year.
9. Non-smokers and non-alcoholics.
10. For female subject is child bearing potential practicing acceptable method of birth control for the duration of the study as judged by Investigator such as Condom, Foams, Jellies,Diaphragm, Intrauterine device and Abstinence.

OR

- is surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. Known history of hypersensitivity to Quetiapine, or related drugs.
2. Requiring medication for any ailment having enzyme-modifying activity in the previous 28 days, prior to dosing day.
3. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
4. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological or psychiatric diseases and bleeding tendency.
5. Participation in a clinical drug study or bioequivalence study within 90 days prior to present study.
6. History of malignancy or other serious diseases.
7. Refusal to abstain from food for at least ten (10.00) hours prior to study drug administration and for at least four (04.00) hours post-dose, in each study period.
8. Any contraindication to blood sampling or difficulty in accessibility of veins.
9. Refusal to abstain from fluid for at least 01.00 hour prior to study drug administration and for at least 01.00 additional hour post-dose, in each study period except about 240 mL of water given during administration of study drug.
10. Refusal to avoid the use of xanthine-containing food or beverages (chocolates,tea, coffee or cola drinks) or fruit juice/grapefruit juice and any alcoholic products for 48.00 hours prior to dosing until the last blood sample collection of last study period.
11. Blood donation within 90 days prior to the commencement of the study.
12. Subjects with positive HIV tests or Hepatitis-B or Hepatitis-C tests.
13. Found positive in breath alcohol test done before check-in for each study period.
14. Found positive in urine test for drugs of abuse done before check-in for each study period.
15. Refusal to abstain from consumption of tobacco products 24.00 hours prior to dosing until the last blood sample collection of last study period.
16. History of problem in swallowing Tablet(s).
17. Female subject, demonstrating positive urine pregnancy test at the time of screening.
18. Female subject, demonstrating positive Serum (ß) Beta- hCG (Human Chorionic Gonadotropin) test before check-in for each study period.
19. Female subject, currently breast feeding or lactating.
20. Female subjects not willing to use acceptable method of contraception from the date of screening until the completion of the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 8 months
  Area Under Curve (AUC)and Cmax Sampling Hours: Pre-dose and at 00.25, 00.50, 00.75, 01.00, 01.25, 01.50, 01.75, 02.00, 02.50, 03.00, 03.50, 04.00, 05.00, 06.00, 08.00, 10.00, 12.00, 24.00, 36.00 and 48.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nirav Gandhi, M.D., Principal Investigator — Accutest Research Lab (I) Pvt. Ltd.
Locations (1):
- Accutest Research Lab (I) Pvt. Ltd., Ahmedabad, Gujarat, India